CLINICAL TRIAL: NCT03204058
Title: Comparative Evaluation of Locally Delivered 1% Metformin and 1.2% Rosuvastatin Gel in Treatment of Intrabony Defects in Chronic Periodontitis Subjects: A Randomized Controlled Clinical Trial
Brief Title: Locally Delivered Metformin & Rosuvastatin for Treatment of Intrabony Defects in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and HOD, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2015-2016DP
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- group 1 (Placebo Comparator): Scaling and root planing (SRP) followed by placebo gel local drug delivery
  Interventions: Drug: Placebos
- group 2 (Active Comparator): SRP followed by 1.2% rosuvastatin (RSV) gel
  Interventions: Drug: Rosuvastatin
- group 3 (Active Comparator): SRP followed by 1% Metformin ( MF) gel
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebos — Oral prophylaxis followed by placement of placebo gel
  Other Names: Inactive drug
  Arms: group 1
Drug: Rosuvastatin — Oral prophylaxis followed by placement of rosuvastatin gel
  Other Names: RSV
  Arms: group 2
Drug: Metformin — Oral prophylaxis followed by placement of metformin gel
  Other Names: MF
  Arms: group 3

SUMMARY:
Metformin (MF), a biguanide group of anti-diabetic drug has been shown to enhance osteoblasts differentiation and inhibit osteoclast differentiation in vitro, thus may exhibit a favourable effect on alveolar bone. Statins are one of the lipid lowering drugs that help in reducing cholesterol levels in the body by specifically inhibiting 3-hydroxy-3-methylglutaryl coenzyme A reductase; which is a rate limiting enzyme for cholesterol synthesis. Rosuvastatin (RSV) have shown to have bone stimulatory and anti-inflammatory effects.Statins are one of the lipid lowering drugs that help in reducing cholesterol levels in the body by specifically inhibiting 3-hydroxy-3-methylglutaryl coenzyme A reductase; which is a rate limiting enzyme for cholesterol synthesis. Rosuvastatin (RSV) and atorvastatin (ATV) have shown to have bone stimulatory and anti-inflammatory effects.. The present study aims to explore the efficacy of 1.2% RSV and 1MF gel as a local drug delivery and redelivery system as an adjunct to scaling and root planing (SRP) for the treatment of intrabony defects.

DETAILED DESCRIPTION:
Metformin (MF), a biguanide group of anti-diabetic drug has been shown to enhance osteoblasts differentiation and inhibit osteoclast differentiation in vitro, thus may exhibit a favourable effect on alveolar bone. Statins are one of the lipid lowering drugs that help in reducing cholesterol levels in the body by specifically inhibiting 3-hydroxy-3-methylglutaryl coenzyme A reductase; which is a rate limiting enzyme for cholesterol synthesis. Rosuvastatin (RSV) have shown to have bone stimulatory and anti-inflammatory effects.Statins are one of the lipid lowering drugs that help in reducing cholesterol levels in the body by specifically inhibiting 3-hydroxy-3-methylglutaryl coenzyme A reductase; which is a rate limiting enzyme for cholesterol synthesis. Rosuvastatin (RSV) and atorvastatin (ATV) have shown to have bone stimulatory and anti-inflammatory effects.. The present study aims to explore the efficacy of 1.2% RSV and 1MF gel as a local drug delivery and redelivery system as an adjunct to scaling and root planing (SRP) for the treatment of intrabony defects.

Methods: Ninety patients with intrabony defects were randomly allocated into three treatment groups: SRP plus placebo gel (group 1), SRP plus 1.2% RSV gel (group 2) and 1% MF gel (group3). Clinical and radiographic parameters were recorded at baseline then after 6 months. The gels were delivered at the respective sites at baseline . Then again all clinical and radiographic parameters were recorded after 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

- All the subjects were systemically healthy subjects with sites having CAL ≥ 3 mm, PPD ≥ 5 mm, vertical bone loss ≥ 3 mm on intraoral periapical radiographs (IOPA) and subjects with no history of periodontal intervention in the last 6 months.

Exclusion Criteria:

patients with systemic diseases like cardiovascular disease diabetes or HIV infection or on medications like corticosteroids which may impede the healing in periodontal tissues.

pregnant/lactating females tobacco users alcoholics patients with unsatisfactory oral hygiene (plaque index greater than 1.5) teeth having gingival recession, caries involving pulp, intrabony defect present interproximally, grade 2/3 mobility Furthermore, patients allergic to Metformin and rosuvastatin or those taking Metformin and rosuvastatin systemically were excluded.

-

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Change in Bone defect fill | baseline, 6 & 12 months
  Assessed in percentage

SECONDARY OUTCOMES:
Change in modified sulcus bleeding index | baseline, 6 & 12 months
  scale 0-3
Change in Plaque index | baseline, 6 & 12 months
  scale 0-3
Change in pocket probing depth | baseline, 6 & 12 months
  measured in mm
Change in clinical attachment level | baseline, 6 & 12 months
  measured in mm
change in intrabony defect depth | baseline, 6 & 12 months
  measured in mm ( Radiograph)